CLINICAL TRIAL: NCT00123630
Title: A Pilot Study of the Treatment of Eosinophilic Esophagitis With Omalizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, John C. Fang, M.D., Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13623
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-03

CONDITIONS: Esophagitis
Keywords: eosinophilic esophagitis; omalizumab
MeSH Terms: conditions — Esophagitis; Eosinophilic Esophagitis | interventions — Omalizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo group
  Interventions: Drug: Placebo
- omalizumab (Experimental): Xolair group
  Interventions: Drug: omalizumab

INTERVENTIONS:
Drug: omalizumab — omalizumab dosed IV based on IgE level and weight every 2 - 4 weeks
  Other Names: Xolair
  Arms: omalizumab
Drug: Placebo — Placebo given IV once every 2-4 weeks based on weight
  Other Names: saline
  Arms: placebo

SUMMARY:
Eosinophilic esophagitis (EE) is an increasingly recognized condition characterized by dysphagia, food impaction or other obstructive esophageal symptoms in children and young adults.

The pathophysiology of EE appears to be an allergy/atopy mediated disease. A personal and family history of allergic diseases (food allergies, atopic dermatitis, asthma, allergic rhinitis or conjunctivitis) has been noted in 62-85% of patients with EE. The rising incidence of EE may be related to the worldwide allergy and asthma epidemic.

Current treatment of EE is directed at decreasing esophageal allergic inflammation. Oral and topical corticosteroids, cromolyn sodium, montelukast and elemental/elimination diets have all been shown to be effective. However, none of these treatments are directed at the specific pathophysiologic mechanism of EE and some have significant side effects.

The shared pathogenetic mechanisms of EE and asthma suggest that therapeutic strategies directed at asthma may also be effective for EE. Specifically those targeted at the allergic immune mechanisms involved with asthma may be effective. Omalizumab is a recently developed anti-IgE antibody that has been shown to decrease the use of inhaled and oral corticosteroids, reduce the frequency of asthma exacerbations, and improve asthma related symptoms in patients with allergic asthma. The objective of the study is to determine the efficacy of omalizumab in the treatment of eosinophilic esophagitis

DETAILED DESCRIPTION:
This is a dual-center double-blind, placebo controlled trial of omalizumab for the treatment of EE. Omalizumab will be dosed depending on the patient's body weight and baseline IgE level. Omalizumab or placebo will be administered subcutaneously every 4 weeks for 16 weeks. At study entry subjects will have EGD with biopsies performed to ensure the diagnosis and obtain tissue for histologic analysis. No dilation will be performed at this time. Baseline validated questionnaires for dysphagia, GERD, and atopy will also be administered. Blood will be drawn for baseline serum testing. Repeat questionnaires and rating of overall symptom improvement will be administered at 4 week intervals for the rest of the study period. At the end of the 16 week period, repeat endoscopy will be performed and biopsies taken. Esophageal dilation may be performed if clinically indicated at this time. Blood will also be drawn for repeat serum testing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 12-60 years of age with EE as defined above
* Serum IgE level 30-700 IU/mL
* Subjects with acceptable medical history, physical exam and laboratory test results
* No history of bleeding diathesis, significant cardiopulmonary disease, or other contraindication to upper endoscopy

Exclusion Criteria:

* Need for esophageal dilation at enrollment due to food impaction or inability to pass endoscope
* Inability of subject to provide informed consent (if ages 18-60), or inability of children (ages 12-17) to provide assent
* History of esophagogastric surgery
* Presence of other esophageal pathology that could account for patients' symptoms including eosinophil infiltration due to gastroesophageal reflux disease (GERD)
* Incarceration
* Pregnancy
* Women of childbearing potential not using the contraception method(s)
* Patients with elevated serum IgE levels for reasons other than atopy
* Patients taking cromolyn sodium or nedocromil sodium within 1 month of visit 1
* Patients taking oral or topical corticosteroids within one month of visit 1
* Patients taking leukotriene receptor inhibitors within one month of visit 1
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Patients with a history of noncompliance to medical regimens or who were considered potentially unreliable
* Use of any other investigational agent in the last 30 days
* Patients with a known hypersensitivity to any ingredient of rhuMAb-E25, study rescue medication
* Patients with Barrett's esophagus will be excluded if found endoscopically or pathologically at biopsy
* Currently treated with omalizumab or treated with omalizumab within the past 6 months.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2005-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Fang, M.D., Principal Investigator — University of Utah HSC
Locations (1):
- University of Utah HSC, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Clayton F, Fang JC, Gleich GJ, Lucendo AJ, Olalla JM, Vinson LA, Lowichik A, Chen X, Emerson L, Cox K, O'Gorman MA, Peterson KA. Eosinophilic esophagitis in adults is associated with IgG4 and not mediated by IgE. Gastroenterology. 2014 Sep;147(3):602-9. doi: 10.1053/j.gastro.2014.05.036. Epub 2014 Jun 4. PMID 24907494

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo 150 to 375 mg is administered SC every 2 or 4 weeks. Because the solution is slightly viscous, the injection may take 5-10 seconds to administer. Doses (mg) and dosing frequency are determined by serum total IgE level (IU/mL), measured before the start of treatment, and body weight (kg).
- Omalizumab: Xolair (Omalizumab)150 to 375 mg is administered SC every 2 or 4 weeks. Because the solution is slightly viscous, the injection may take 5-10 seconds to administer. Doses (mg) and dosing frequency are determined by serum total IgE level (IU/mL), measured before the start of treatment, and body weight (kg).
Period: Overall Study
Arm/Group | Placebo | Omalizumab
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omalizumab | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6) | 32 (12) | 30 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Eosinophil Numbers Per High Power Field Proximally and Distally Between Baseline and Post-treatment and Between Both Groups
Time Frame: 16 weeks
Population: The analysis was per protocol. There were no subjects who were withdrawn or lost to follow-up in this study.
Measure: Number; unit: perecentage of eos per high power field
Arm/Group | Placebo | Omalizumab
Number analyzed (Participants) | 15 | 15
perecentage of eos per high power field | 0.6 | -7.5
Statistical Analysis 1: Comparison: Placebo vs Omalizumab; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Placebo | Omalizumab
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
small numbers enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less